CLINICAL TRIAL: NCT05074459
Title: Interventional, Randomized, Double-blind, Parallel-group, Healthy Subject, Single Dose Study Investigating the Safety, Tolerability, and Pharmacokinetic Properties of Eptinezumab Manufactured Using Two Different Cell Lines
Brief Title: A Study in Healthy Adults Investigating Eptinezumab Produced by 2 Different Manufacturing Cell Lines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19889A
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eptinezumab Mammalian Cell Line (Experimental): Participants will receive a single intravenous (IV) infusion of eptinezumab mammalian cell line on Day 1.
  Interventions: Drug: Eptinezumab Mammalian Cell Line
- Eptinezumab Yeast Cell Line (Active Comparator): Participants will receive a single IV infusion of eptinezumab yeast cell line on Day 1.
  Interventions: Drug: Eptinezumab Yeast Cell Line

INTERVENTIONS:
Drug: Eptinezumab Mammalian Cell Line — Concentrate for solution for IV infusion
  Arms: Eptinezumab Mammalian Cell Line
Drug: Eptinezumab Yeast Cell Line — Concentrate for solution for IV infusion
  Arms: Eptinezumab Yeast Cell Line

SUMMARY:
Eptinezumab is a preventive treatment for migraine. The drug is made from a process that currently uses yeast cells for production of the drug. The trial researchers want to test whether using a new production cell line to make eptinezumab will affect the way the drug behaves in the body. To do this, the researchers will give a single dose of eptinezumab to healthy participants. Some of the participants will get eptinezumab that has been made from yeast cells. Others will get eptinezumab made with the new cell line.

ELIGIBILITY:
Key Inclusion Criteria:

* The participant has a body weight ≥50 and ≤100 kilograms (kg).
* The participant has a body mass index (BMI) ≥18.5 and ≤30 kg/meter (m^2) at the screening visit and at the baseline visit.
* The participant has a resting supine pulse ≥45 and ≤100 beats per minute (bpm) at the screening visit and at the baseline visit.
* The participant has a resting supine systolic blood pressure ≥91 and ≤140 millimeters of mercury (mmHg) and a resting supine diastolic blood pressure ≥51 and ≤85 mmHg at the screening visit and at the baseline visit.
* The participant is, in the opinion of the investigator, generally healthy based on medical history, a physical examination, vital signs, an electrocardiogram (ECG), and the results of the clinical chemistry, haematology, urinalysis, serology, and other laboratory tests.

Key Exclusion Criteria:

* The participant has taken disallowed medication <1 week prior to the dose of investigational medicinal product (IMP) or <5 half-lives prior to the screening visit for any medication taken.
* The participant has taken any IMP <3 months or <5 half-lives (whichever is longer) prior to the first dose of IMP.
* The participant has or has had any clinically significant immunological, cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, haematological, dermatological, venereal, neurological, or psychiatric disease or other major disorder.
* The participant has been dosed with a monoclonal antibody (mAb) ≤6 months prior to the screening visit.
* The participant is a smoker or uses other nicotine-containing products (for example, snuff, nicotine patches, nicotine chewing gum, mock cigarettes, inhalers). Ex-smokers must have ceased smoking >3 months prior to the screening visit.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Area Under the Eptinezumab Plasma Concentration-Time Curve (AUC) From Zero to Infinity (AUC0-inf) | Day 1 (pre-dose up to 12 hours after the end of the infusion) up to Day 112 (after the end of the infusion), and at the follow-up visit Day 140

SECONDARY OUTCOMES:
Percent Extrapolated AUC of Total AUC0-inf (AUC%extr) | Day 1 (pre-dose up to 12 hours after the end of the infusion) up to Day 112 (after the end of the infusion), and at the follow-up visit Day 140
Maximal Observed Plasma Concentration (Cmax) | Day 1 (pre-dose up to 12 hours after the end of the infusion) up to Day 112 (after the end of the infusion), and at the follow-up visit Day 140
Area Under the Plasma Concentration-Time Curve From Zero to Time t (AUC0-t) | Day 1 (pre-dose up to 12 hours after the end of the infusion) up to Day 112 (after the end of the infusion), and at the follow-up visit Day 140
Apparent Terminal Elimination Half-Life (t½) | Day 1 (pre-dose up to 12 hours after the end of the infusion) up to Day 112 (after the end of the infusion), and at the follow-up visit Day 140
Systemic Clearance (CL), Defined as Dose/AUC0-inf | Day 1 (pre-dose up to 12 hours after the end of the infusion) up to Day 112 (after the end of the infusion), and at the follow-up visit Day 140
Apparent Volume of Distribution (Vz) | Day 1 (pre-dose up to 12 hours after the end of the infusion) up to Day 112 (after the end of the infusion), and at the follow-up visit Day 140

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — H. Lundbeck A/S
Locations (2):
- United States (2):
  - Labcorp Clinical Research Unit, Inc., Daytona Beach, Florida
  - Labcorp Clinical Research Unit, Inc., Madison, Wisconsin